CLINICAL TRIAL: NCT04046016
Title: A Phase 0 Study to Investigate Biodistribution and Target Tissue Distribution Using Whole-body PET Scan After Oral Administration of Therapeutic Dose of Liporaxel Solution and Microdose of 18F-labeled Liporaxel in Patients With Solid Tumor
Brief Title: A Study Using Whole-body PET After Oral Microdose of 18F-labeled Liporaxel in Patients With Solid Tumor
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Howard Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHP107_Bioimaging
Record Dates: First submitted 2019-05-17; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects (Experimental): A total of two subjects were enrolled. Those are breast cancer patients.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Liporaxel and microdose 18F-Liporaxel administration study was conducted in two breast cancer patients. Therapeutic dose of Liporaxel was 200 mg/m2 and 18F-Liporaxel was 0.98-2.9 μg (185-555 MBq).
  Other Names: Liporaxel

SUMMARY:
An open-label, single oral dose of therapeutic Liporaxel and microdose 18F-Liporaxel administration study was conducted in two breast cancer patients. Therapeutic dose of Liporaxel was 200 mg/m2 and 18F-Liporaxel was 0.98-2.9 μg (185-555 MBq).

DETAILED DESCRIPTION:
The subject should be diagnosed as solid cancer on histopathology or cytology and should be more than 19 years old. Patients with progressed, metastatic, or recurrent disease despite standard therapies for solid tumors were included. The disease had to be measurable according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The Eastern Cooperative Oncology Group (ECOG) performance status should be less than 2 and the predicted survival time should be more than 12 weeks. Those who were not able to take the oral medication or who had an operation that could lead to abnormal bile acid secretion were excluded. Patients with a history of adverse reactions and allergic reactions to paclitaxel or paclitaxel-like substances (e.g., taxol) were also excluded. Patients who are taking P-glycoprotein inducers or inhibitors or drugs which is known to exist drug-drug interaction with paclitaxel (e.g., cyclosporine A, ketoconazole, rifampicin, clarithromycin) were excluded. Patients with a neutrophil count less than 1,500 cell/mm3, platelet count less than 100,000 cells/mm3, and with infectious diseases at the beginning of the study were excluded.

Subjects eligible for the inclusion/exclusion criteria were orally administered Liporaxel solution 300 mg containing a microdose amount of 18F-Liporaxel on Visit 1. At 0, 2, 4, 8, 10 h post-dose, whole body PET/CT imaging (head-to-thigh) were obtained. Visit 2, 3, and 4 were taken 1, 2, and 3 weeks after Visit 1, respectively. For each visit, the adverse events, vital sign, physical examination, and clinical laboratory test results were evaluated and then therapeutic dose of Liporaxel was administered. Five weeks after Visit 1, the subject self-administered Liporaxel and adverse events and comedication were followed up by phone. At Visit 6, eight weeks after Visit 1, RECIST measurements were made with contrast-enhanced CT with safety evaluation. Tumor response was assessed to determine whether the study could be completed. If the tumor response was progression, the study was to be terminated. If stable disease, subject started a new cycle starting from Visit 6, and decided to evaluate tumor response with CT scan every eight week based on Visit 6. If the subject did not adequately recover from the hematologic and non-hematologic toxicities of Liporaxel during the entire study, the doses could be delated for up to two weeks at the discretion of the investigator. Exclusion was made in cases exceeding two weeks.

ELIGIBILITY:
Inclusion criteria:

1. The subject should be diagnosed as solid cancer on histopathology or cytology and should be more than 19 years old.
2. Patients with progressed, metastatic, or recurrent disease despite standard therapies for solid tumors were included.
3. The disease had to be measurable according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
4. The Eastern Cooperative Oncology Group (ECOG) performance status should be less than 2 and the predicted survival time should be more than 12 weeks.

Exclusion criteria:

1. Those who were not able to take the oral medication or who had an operation that could lead to abnormal bile acid secretion were excluded.
2. Patients with a history of adverse reactions and allergic reactions to paclitaxel or paclitaxel-like substances (e.g., taxol) were also excluded.
3. Patients who are taking P-glycoprotein inducers or inhibitors or drugs which is known to exist drug-drug interaction with paclitaxel (e.g., cyclosporine A, ketoconazole, rifampicin, clarithromycin) were excluded.
4. Patients with a neutrophil count less than 1,500 cell/mm3, platelet count less than 100,000 cells/mm3, and with infectious diseases at the beginning of the study were excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Cmax | pre-dose, 2, 4, 6, 8, 10 hours after post-dose
  Plasma paclitaxel peak concentration
AUClast | pre-dose, 2, 4, 6, 8, 10 hours after post-dose
  Plasma paclitaxel area under the time-concentration curve until the last measurable time point

CONTACTS AND LOCATIONS:
Overall Officials: Howard Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyounggi, South Korea

IPD SHARING:
Plan to Share IPD: No